CLINICAL TRIAL: NCT00002163
Title: A Phase III, Randomized, Double-Blind, Multicentre Study to Evaluate the Safety and Efficacy of 1592U89 in Patients With AIDS Dementia Complex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 238B; CNAB 3001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: AIDS Dementia Complex; HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS Dementia Complex; Antiviral Agents; abacavir
MeSH Terms: conditions — AIDS Dementia Complex; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
To evaluate the benefit of adding 1592U89 to current antiretroviral therapies for AIDS dementia complex and to assess the safety and tolerance of the treatment regimens.

DETAILED DESCRIPTION:
Patients must be on stable antiretroviral treatment for at least 6 weeks prior to study entry and will then be stratified depending on whether their regimen contains zidovudine (ZDV). Each stratum will be randomized separately to receive 1592U89 or placebo for 12 weeks. For the subsequent 40 weeks, open-label 1592U89 will be offered.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* Evidence of HIV - associated dementia.
* Been on stable antiretroviral treatment for a minimum of 6 weeks prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Debilitated as a result of their HIV disease, associated illness or therapies who the investigator determines will not be able to complete the 12 week randomized dosing period.
* Memorial Sloan-Kettering (MSK) score of >= 3 for dementia.
* Confounding neurological diseases which may interfere with interpretation of neurological and neurophysical assessments.
* Malabsorption syndrome or other gastrointestinal dysfunction which renders them unable to take oral medication.
* Chronic diseases such as diabetes, congestive heart failure, cardiomyopathy, other cardiac dysfunctions, etc., which in the investigator's opinion would compromise the safety of the patient.
* Symptomatic AIDS-defining opportunistic infection not responsive to therapy.

Concurrent Medication:

Excluded:

* Treatment with cytotoxic chemotherapeutic agents within the first 12 weeks of the study.
* Treatment with nerve growth factor within the first 12 weeks of study.
* The use of narcotic analgesics, sedatives, benzodiazepines, antidepressants, anti-psychotic agents and other psychoactive drugs which would interfere with the assessment of the neurological and neurophysical status of the patient.
* Use of stavudine (d4T) during the first 12 weeks of the study.
* Immunomodulating agents (except GM/G-CSF or epoietin).
* Psychoactive drugs (at the investigator's discretion).

Concurrent Treatment:

Excluded:

* Treatment with radiation therapy within the first 12 weeks of the study.

NOTE:

* With the exception of local treatment for Kaposi's sarcoma.

Patients with any of the following prior conditions are excluded:

* Previous neurological disease unrelated to HIV infection.
* History of clinically apparent hepatitis within the last 6 months.
* History of clinically apparent pancreatitis in the last 6 months.

Prior Medication:

Excluded:

* Treatment with cytotoxic chemotherapeutic agents within 1 month of entry.
* Participation in investigational antiretroviral trials within the past 3 months.
* HIV vaccine within the past 3 months.
* Treatment with immunomodulating agents such as systemic corticosteroids, interleukins, thalidomide, anticytokine agents, anti-oxidants or interferons within 1 month of study entry.
* Nerve growth factor.

Prior Treatment:

Excluded:

* Treatment with radiation therapy within 1 month of entry.

NOTE:

* With the exception of local treatment for Kaposi's sarcoma.

Risk Behavior:

Excluded:

Current alcohol or illicit drug use which may interfere with the patient's ability to comply with the study protocol.

Required:

* Stable antiretroviral treatment that has been ongoing for a minimum of 6 weeks prior to study entry, may or may not include ZDV.

Required:

* Stable antiretroviral treatment for a minimum of 6 weeks prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - HIV Neurobehavioral Research Ctr, San Diego, California
  - San Francisco Gen Hosp, San Francisco, California
  - Johns Hopkins Univ School of Medicine, Baltimore, Maryland
  - Washington Univ Med Ctr, St Louis, Missouri
  - Mount Sinai Med Ctr, New York, New York
  - Columbia Univ / Sergievsky Ctr, New York, New York
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina
- Canada (2):
  - Univ of Manitoba / Faculty of Medicine, Winnipeg, Manitoba
  - Wellesley Hosp, Toronto, Ontario

REFERENCES:
- [Background] Lanier ER, Sturge G, McClernon D, Brown S, Halman M, Sacktor N, McArthur J, Atkinson JH, Clifford D, Price RW, Simpson D, Torres G, Catalan J, Marder K, Power C, Hall C, Romero C, Brew B. HIV-1 reverse transcriptase sequence in plasma and cerebrospinal fluid of patients with AIDS dementia complex treated with Abacavir. AIDS. 2001 Apr 13;15(6):747-51. doi: 10.1097/00002030-200104130-00010. PMID 11371689